CLINICAL TRIAL: NCT06437964
Title: The Use of Prophylactic Antibiotics in the Endoscopic Secondary Prevention of Cirrhotic Patients With Gastroesophageal Variceal Bleeding
Brief Title: Prophylactic Antibiotics in Endoscopic Secondary Prevention of Gastroesophageal Variceal Bleeding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0629
Record Dates: First submitted 2024-05-26; First posted 2024-05-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Cirrhosis, Liver; Hypertension, Portal; Variceal Hemorrhage
Keywords: Gastroesophageal Variceal Bleeding; Endoscopic Secondary Prevention; Prophylactic Antibiotics
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prophylactic antibiotics (Active Comparator): Intravenous infusion of 1.0g-2.0g ceftriaxone before endoscopic therapy
  Interventions: Drug: Prophylactic Antibiotics
- No prophylactic antibiotics (Experimental): No use of prophylactic antibiotics before endoscopic therapy
  Interventions: Other: No use of prophylactic antibiotics

INTERVENTIONS:
Other: No use of prophylactic antibiotics — In the endoscopic secondary prevention of cirrhotic patients with gastroesophageal variceal bleeding, do not use any antibiotics before the endoscopic operation.
  Arms: No prophylactic antibiotics
Drug: Prophylactic Antibiotics — Intravenous infusion of 1.0g-2.0g ceftriaxone before endoscopic therapy
  Arms: Prophylactic antibiotics

SUMMARY:
Whether prophylactic antibiotics should be administered in the endoscopic secondary prevention of GVB or not is unclear. In this non-inferiority trial, we are aimed to evaluate whether prophylactic antibiotics are essential in the endoscopic secondary prevention of cirrhotic patients with gastroesophageal variceal bleeding.

DETAILED DESCRIPTION:
Prophylactic antibiotics like third-generation cephalosporin is recommended for acute gastroesophageal variceal bleeding (GVB). Endoscopic sequential therapy is an option in the secondary prevention of acute gastroesophageal variceal bleeding (GVB). However, the value of prophylactic antibiotics in the endoscopic secondary prevention of GVB is still unclear. It's assumed that the procedure of needle puncture under endoscopy will cause iatrogenic variceal bleeding. Besides, the surface of intraluminal varices is nonsterile, and injection of sclerosing agent or tissue adhesive will put patients at a risk of bacteremia. As a result, it's rational to use antibiotics prophylactically in the endoscopic sequential therapy of GVB. While giving antibiotics in all patients might cause abuse of antibiotics. In clinical practice now, the prophylactic administration of antibiotics is quite subjective. We observe that quite a lot of cirrhotic patients had no infection after endoscopic secondary prevention for gastroesophageal variceal bleeding, even they have not been administered prophylactic antibiotics. In this non-inferiority trial, we are aimed to evaluate whether no value of prophylactic antibiotics will increase the postoperative infection or not, in the endoscopic secondary prevention of cirrhotic patients with gastroesophageal variceal bleeding.

ELIGIBILITY:
Inclusion Criteria:

Cirrhotic patients having a history of gastroesophageal variceal bleeding are readmitted for endoscopic secondary prevention.

Exclusion Criteria:

1. Age <18, or ≥81.
2. The patient is unwilling to sign the informed consent form.
3. Allergy to cephalosporin.
4. Have granulocyte deficiency (neutrophil count ≤ 0.5 * 10 ^ 9/L, or white blood cell count ≤ 1.0 * 10 ^ 9/L) before the endoscopic operation.
5. Already have infection or fever (body temperature > 37.5 ℃) before signing the informed consent form.

Withdraw Criteria:

1. The patient turned back after signing the consent, and before the endoscopic operation.
2. Have fever (body temperature > 37.5 ℃) after signing the consent, and before the endoscopic operation.
3. Transferred to other department for additional treatment after the endoscopic operation (Surgical department for malignant tumor, Interventional radiology department for splenic embolism or transjugular intrahepatic portosystemic shunt, etc.).
4. The patient suffered massive bleeding during the endoscopy, and cephalosporin was given immediately after being sent back to the ward.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Actual)
Dates: Start 2024-05-25 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-02-10 (Estimated)

PRIMARY OUTCOMES:
Postoperative fever | From the date of endoscopic operation (after the endoscopy) until the date of hospital discharge, assessed up to 7 days.
  Have fever (>37.5℃) in hospital afer the endoscopic operation

SECONDARY OUTCOMES:
Postoperative 4-week rebleeding | Within 4 weeks since the endoscopic operation
  Have gastroesophageal variceal bleeding within 4 weeks after the endoscopic operation
Additional use of antibiotics | From the date of endoscopic operation (after the endoscopy) until the date of hospital discharge, assessed up to 7 days.
  Received additional antibiotics after the endoscopic operation
Postoperative hospital stays | From the date of endoscopic operation until the date of hospital discharge, assessed up to 7 days.
  Hospital stay (days) after the endoscopic operation

CONTACTS AND LOCATIONS:
Overall Officials: Meng Xue, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, ZhejiangUniversity
Locations (1):
- The 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No